CLINICAL TRIAL: NCT02093494
Title: A Randomized, Open Label Study to Evaluate the Effectiveness of the MMT Initial Specimen Diversion Device in Reducing Blood Culture Contamination Compared to Laboratory Standard Procedures When Collected Through Peripheral Intravenous Catheters (PIVC)
Brief Title: Study to Evaluate the Effectiveness of the Initial Specimen Diversion Device When Collected Through Peripheral Intravenous Catheters
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Magnolia Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMT1303
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Septicemia
Keywords: Septicemia; Blood culture; Contamination
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial Specimen Diversion Device (ISDD) (Experimental): The ISDD will be used to collect the blood culture.
  Interventions: Device: Initial Specimen Diversion Device (ISDD)
- Lab standard practice (LSP) (Active Comparator): The ISDD will not be used to collect the blood culture. Standard blood culture specimen collection kits will be utilized.
  Interventions: Procedure: Lab standard practice (LSP); Device: Peripheral Intravenous Catheters (PIVC)

INTERVENTIONS:
Device: Initial Specimen Diversion Device (ISDD)
  Arms: Initial Specimen Diversion Device (ISDD)
Procedure: Lab standard practice (LSP)
  Arms: Lab standard practice (LSP)
Device: Peripheral Intravenous Catheters (PIVC)
  Arms: Lab standard practice (LSP)

SUMMARY:
This is a randomized, open label study to evaluate the Initial Specimen Diversion Device (ISDD) in reducing the contamination rate in blood culture analysis. Blood culture data will be derived from inpatient and/or outpatient settings in a variety of hospital departments (e.g. ER, surgical, medical, etc.). Only samples that are collected via PIVC's may be included in this study. The ISDD will be compared to current laboratory practices for the collection of blood for culture purposes. Laboratory Standard Procedures (LSP) is defined as collection of venipuncture blood for culture without an initial diversion method to divert and sequester potential blood contaminants.

ELIGIBILITY:
Inclusion Criteria:

* Adults >19 years old

Exclusion Criteria:

* Not a good candidates for direct-to-media (DTM) technique

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the rate of blood culture contamination using the Initial Specimen Diversion Device (ISDD) compared to Laboratory Standard Procedures (LSP) when collected through PIVC | Baseline

SECONDARY OUTCOMES:
Evaluate the occurrence of any adverse device effects | Baseline
  As the device under study enhances the blood diversion procedure during blood culture collection, and is part of standard blood collection standards, adverse device effects are not expected as a result of use of this device. Any issues with the function of the device will be reported by the phlebotomist on a device incident form. The sponsor will maintain these reports in a database. As this is a commercially available device, medical device reporting shall be performed in accordance with 21 CFR 803, as applicable.

OTHER OUTCOMES:
Evaluate the contamination rates, taking into account the confounding effects of blood draw setting and departure from direct-to-media (DTM) technique | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Richard Patton, M.D., Study Director — Magnolia Medical Technologies, Inc.
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States